CLINICAL TRIAL: NCT00359814
Title: Conversion Study to Optimize Immunosuppressive Regimen by Exchange of Azathioprine by Mycophenolatmofetile and Cyclosporine A Dose Reduction for Patients After Heart Transplantation in Lon-Term
Brief Title: Exchange of Azathioprine by Mycophenolatmofetile and Cyclosporine A Dose Reduction After Heart Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Dr. med. Christoph Bara, Clinic for Cardiothoracic, Transplantation and Vascular Surgery, HannoverMS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KKS-95/2004
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Heart Transplantation
Keywords: Cyclosporine; renal insufficiency, chronic; long-term care
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Mycophenolic Acid; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Azathioprine administration: was stopped at day 0; Mycophenolatmofetile administration: was started with 250 mg/daily at day 1, the start dose was increased about 250 mg/daily every week till 2 g/daily; Cyclosporin A reduction: Cyclosporin A trough level reduction started after week 8. The new target range was 50 to 90 ng/ml
  Interventions: Drug: Mycophenolatmofetile; Drug: Cyclosporin A

INTERVENTIONS:
Drug: Mycophenolatmofetile — Mycophenolatmofetile administration: was started with 250 mg/daily at day 1, the start dose was increased about 250 mg/daily every week till 2 g/daily
  Other Names: MMF; CellCept
Drug: Cyclosporin A — Cyclosporin A reduction: Cyclosporin A trough level reduction started after week 8. The new target range was 50 to 90 ng/ml
  Other Names: Sandimmun optoral

SUMMARY:
The purpose of this study is to improve or save renal function by optimizing the immunosuppressive regimen by reducing the Cyclosporine A dose and the exchange of Azathioprine by Mycophenolatmofetile, which is an effective immunosuppressive agent and will minimize the risk of acute rejection episodes.

DETAILED DESCRIPTION:
The decrease of quality of life in patients after heart transplantation in the long-term is determined by an increasing incidence of transplant vasculopathy and by immunosuppression-related side effects.Long-term administration of calcineurin inhibitors is associated with chronic nephrotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Current immunosuppressive regimen: Cyclosporine A, Azathioprine and corticosteroids for at least 12 month
* Heart transplantation above 3 years dated back
* Serum creatinine < 3,5 mg/dl (310 µmol/l) and BUN < 150 mg/dl
* Cyclosporine A blood level between 50 and 250 ng/ml during the last 12 month

Exclusion Criteria:

* Carcinoma within the last 3 years
* Acute rejection episodes during the last 6 month
* Infection requiring therapeutic intervention
* Hepatitis B, Hepatitis C or HIV infection
* WBC < 3000/µl, haemoglobin < 9g/dl, platelets < 70.000/µl
* Florid gastrointestinal ulcer
* Haemodialysis within the last 4 weeks before study entry
* Pregnancy / lactation
* Administration of other immunosuppressive agents than prescribed
* Mycophenolatmofetile incompatibility

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Renal function evaluated by serum creatinine at month 12 and month 24 | month 12 and month 24

SECONDARY OUTCOMES:
acute rejection episodes, gastrointestinal disorders and other adverse events at month 12 and month 24 | month 12 and month 24
Cardiovascular risk factors at month 12 and month 24 | month 12 and month 24
Quality of life assessed by the SF36, spiroergometry, concomitant medication at month 12 and month 24 | month 12 and month 24

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Bara, Dr. med., Study Director — Hannover Medical School, Department of Thoracic and Cardiovascular Surgery
Locations (1):
- Hannover Medical School, Department of Thoracic and Cardiovascular Surgery, Hanover, Germany